CLINICAL TRIAL: NCT00870064
Title: The Treatment of Type I Open Fractures in Pediatrics: Evaluating the Necessity of Formal Irrigation and Debridement
Brief Title: The Treatment of Type I Open Fractures in Pediatrics
Acronym: PROOF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other); University of Mississippi Medical Center (Other); MultiCare Mary Bridge Children's Hospital & Health Center (Other); Yale New Haven Health System Center for Healthcare Solutions (Other); University of New Mexico Carrie Tingley Hospital (Unknown); IWK Health Centre (Other); Phoenix Children's Hospital (Other); Children's Hospital Colorado (Other); Nationwide Children's Hospital (Other); Morristown Medical Center (Other); NYUMC-Hospital for Joint Diseases (Unknown); Children's Medical Center Dallas (Other); Johns Hopkins University (Other); Orthopaedic Institute for Children (Other); Children's Hospital Los Angeles (Other); St. Christopher's Hospital for Children (Other); Children's Hospital of Orange County (Other)
Responsible Party: Principal Investigator, Joseph Janicki, MD, Assistant Professor of Pediatrics, Northwestern University Feinberg School of Medicine, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-13763
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-01

CONDITIONS: Fractures, Open
Keywords: Surgical Procedures, Operative; Fractures, Open; Fracture Fixation
MeSH Terms: conditions — Fractures, Open

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Formal Operative Treatment (Other): Children randomized to the formal operative management arm will be taken to the Operating Room within 24 hours for irrigation and debridement and appropriate bone management.
  Interventions: Procedure: Formal Operative Treatment
- Emergency Department Treatment (Other): Children in the Emergency Department Treatment arm will have a washout in the emergency room under conscious sedation, a closed reduction and home antibiotics.
  Interventions: Procedure: Emergency Department Treatment

INTERVENTIONS:
Procedure: Formal Operative Treatment — Children randomized to the OR arm will be taken to the OR within 24 hours for irrigation and debridement and appropriate bone management.
  Arms: Formal Operative Treatment
Procedure: Emergency Department Treatment — Children in the ED arm will have a washout in the emergency room under conscious sedation, a closed reduction and home antibiotics.
  Arms: Emergency Department Treatment

SUMMARY:
Open fractures are frequently encountered in orthopaedics. Treatment usually calls for a formal, operative procedure in which the bone is exposed, foreign tissue is debrided and the wound is irrigated. While this is the current standard of care, not all open fractures are equal. In retrospective studies, centers are reporting less aggressive operative management for open fractures may result in equal results without the time and expense of the operative theater. The investigators propose a prospective, randomized trial of children with type I open fractures to evaluate whether formal operative treatment is necessary. The investigators' hypothesis is that minor open fractures can be safely treated in the emergency room with irrigation, closed reduction and home antibiotics without an increased risk of infection or other complications. Children who meet the study criteria will be randomized into two treatment arms - formal operative management (OR) and emergency department (ED) management. Outcomes from each group will be evaluated and compared, including rate of infection, number of return visits to the operating room, time to union, and other complications.

DETAILED DESCRIPTION:
Fractures in which bone has been exposed to the outside world through an associated skin injury, known as open fractures, are frequently encountered in orthopaedics. Traditionally, treatment calls for a formal, operative treatment in which the bone is exposed, foreign tissue is debrided and the wound is irrigated. The bone itself, depending on the age of the patient, fracture location and stability is then treated by the appropriate method of casting or internal fixation. However, while this is the current standard of care for all open fractures, not all open fractures are the same and can differ in terms of the bone involved, energy causing the injury and the skeletal maturity of the patient. Children, for example, have a thick periosteum which may diminish the rate of infection and decrease the time to healing. In addition, the protocol of operative debridement was introduced at the same time as widespread antibiotic use. It is not known whether the mechanical operative management or antibiotic use has resulted in improved outcomes. In retrospective studies, centers are reporting emergency department management alone may result in equal results without the time and expense of the operative theater.

The investigators propose a prospective, randomized trial of children with type I open fractures to evaluate whether formal operative treatment is necessary. The investigators hypothesize that minor open fractures in children can be safely treated in the emergency room with irrigation, closed reduction and home antibiotics without an increased risk of infection or other complications. If the inclusion criteria is met and informed consent is obtained, children will be randomized into two treatment arms - formal operative management (OR) and emergency department (ED) management. Children randomized to the OR arm will be taken to the OR within 24 hours for irrigation and debridement and appropriate bone management. Children in the ED arm will have a washout in the emergency room under conscious sedation, a closed reduction and home antibiotics. Both wounds will be examined at interval follow up periods for signs of infection. Outcomes evaluated will include the rate of infection, the number of return visits to the operating room, the time to bone healing, and other complications. This is a pilot study with the plan of eventually being a multicenter study evaluating open fracture care in children.

ELIGIBILITY:
Inclusion Criteria:

* open fracture amenable to treatment by closed reduction
* low energy mechanism of injury (e.g., falls from less than 10 feet, bicycle accidents)
* wound less than 1cm in length and the bone not visualized through the skin

Exclusion Criteria:

* open fracture not amenable to treatment by closed reduction
* open fracture that would typically require operative reduction and fixation
* high energy mechanism of injury (e.g., struck by vehicle, motor vehicle accidents, fall from height greater than 10 feet)
* wound greater than 1cm in length
* gross contamination of wound
* open fractures involving hands or feet (the current standard of care to treat open injuries involving hands or feet is only emergency room management)

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2010-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of infection | 2 weeks
  1. Do patients with type one open fractures treated in the emergency department with irrigation have a non-inferior rate of infections compared to those treated in the operating room with formal irrigation and debridement? The response variable will be the presence of an infection in children with open fractures.

SECONDARY OUTCOMES:
Time to bone healing | 24 weeks
  2. Do patients with type I open fractures who are treated nonoperatively have a non-inferior time to bone healing when compared to those treated operatively? The response variable will be time to clinical and radiographic fracture healing.
Return visits to OR | 24 weeks
  Number of return visits to the operating room

CONTACTS AND LOCATIONS:
Overall Officials: Joseph (Jay) A Janicki, MD, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Yang EC, Eisler J. Treatment of isolated type I open fractures: is emergent operative debridement necessary? Clin Orthop Relat Res. 2003 May;(410):289-94. doi: 10.1097/01.blo.0000063795.32430.4c. PMID 12771843
- [Background] Iobst CA, Tidwell MA, King WF. Nonoperative management of pediatric type I open fractures. J Pediatr Orthop. 2005 Jul-Aug;25(4):513-7. doi: 10.1097/01.bpo.0000158779.45226.74. PMID 15958906
- [Background] Doak J, Ferrick M. Nonoperative management of pediatric grade 1 open fractures with less than a 24-hour admission. J Pediatr Orthop. 2009 Jan-Feb;29(1):49-51. doi: 10.1097/BPO.0b013e3181901c66. PMID 19098646
- [Background] Gustilo RB, Anderson JT. Prevention of infection in the treatment of one thousand and twenty-five open fractures of long bones: retrospective and prospective analyses. J Bone Joint Surg Am. 1976 Jun;58(4):453-8. PMID 773941
- [Background] Grimard G, Naudie D, Laberge LC, Hamdy RC. Open fractures of the tibia in children. Clin Orthop Relat Res. 1996 Nov;(332):62-70. doi: 10.1097/00003086-199611000-00009. PMID 8913146
- [Background] Haasbeek JF, Cole WG. Open fractures of the arm in children. J Bone Joint Surg Br. 1995 Jul;77(4):576-81. PMID 7615601
- [Background] Skaggs DL, Kautz SM, Kay RM, Tolo VT. Effect of delay of surgical treatment on rate of infection in open fractures in children. J Pediatr Orthop. 2000 Jan-Feb;20(1):19-22. PMID 10641682
- [Background] Jones BG, Duncan RD. Open tibial fractures in children under 13 years of age--10 years experience. Injury. 2003 Oct;34(10):776-80. doi: 10.1016/s0020-1383(03)00031-7. PMID 14519359
- [Background] Jones IE, Williams SM, Dow N, Goulding A. How many children remain fracture-free during growth? a longitudinal study of children and adolescents participating in the Dunedin Multidisciplinary Health and Development Study. Osteoporos Int. 2002 Dec;13(12):990-5. doi: 10.1007/s001980200137. PMID 12459942
- See also: Center for Disease Control. (12 April 2024). Surgical Site Infection. In Center for Disease Control and Prevention. Retrieved August 28, 2024 — https://www.cdc.gov/infection-control/hcp/surgical-site-infection/index.html